CLINICAL TRIAL: NCT03745768
Title: Intermittent Theta Burst Stimulation to Relieve Depression and Concurrent Executive Function Impairment in Older Adults: A Randomized Controlled Study
Brief Title: iTBS Study for Depression (Randomized)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201803023
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Executive Dysfunction; Depression
Keywords: depression; executive dysfunction; transcranial magnetic stimulation; intermittent theta burst stimulation; neuromodulation; older adults; geriatrics
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial testing iTBS versus sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active iTBS Treatment (Experimental): Participants received Intermittent theta burst stimulation to the dorsolateral prefrontal cortex for 6 weeks
  Interventions: Device: Intermittent Theta Burst Stimulation
- Sham Stimulation (Sham Comparator): Participants received Sham stimulation to the dorsolateral prefrontal cortex for 6 weeks.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — Intermittent theta burst stimulation delivered to the dorsolateral prefrontal cortex on the left and right sides of the brain for 6 weeks.
  Arms: Active iTBS Treatment
Device: sham stimulation — Sham stimulation delivered to the dorsolateral prefrontal cortex on the left and right sides of the brain for 6 weeks.
  Arms: Sham Stimulation

SUMMARY:
Executive function deficits are common in late life depression (LLD) and are associated with resistance to antidepressants, poor quality of life, considerable disability and increased suicidal risk. This study uses a novel type of Transcranial Magnetic Stimulation called intermittent Theta Burst Stimulation (iTBS). iTBS delivers high frequency (50Hz) magnetic pulses in "bursts" of 3 stimuli. It is posited that this intervention induces plasticity in the human cortex. Theoretical and empirical evidence from research studies informs that iTBS can improve depression and executive deficits, however, this has not been examined in older adults.

This project examines iTBS's ability to improve depression and executive impairment in LLD. It also tests the effects of iTBS on brain connectivity within the Cognitive Control Network (CCN). This study will enhance understanding of LLD, providing critical pilot data to develop future randomized controlled clinical trials.

Both active and sham interventions are administered sequentially to the left and right dorso-lateral prefrontal cortex. The total stimulation time is about 7 minutes. These interventions are administered for 6 weeks (Monday-Friday). 20 subjects will be randomized. Changes in mood from baseline to the end of study are measured with the Montgomery-Asberg Depression Rating Scale. Executive function at baseline and end of study are evaluated with the National Institutes of Health Toolbox executive domain battery. Safety assessments include: the 21 item Scale for suicidal ideation SSI. The frequency, intensity and burden of side effects rating (FIBSER) and the Altman Self Rating Mania scale (ASRM). Ancillary depression measures include the Quick Inventory of Depressive Symptoms (QIDS) and the Clinical Global Impression of Improvement scale.

Subjects undergo functional Magnetic Resonance Imaging (fMRI) before and after the study interventions to test the effects of iTBS on the brain's functional connectivity.

This research will provide meaningful information about the effects of iTBS on mood and executive function in older adults as well as information regarding its effects on brain function. Results of this pilot study will inform a grant submission and allow investigators to calculate power for a definitive randomized controlled clinical trial to test the efficacy of iTBS versus placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 - 85 years old
2. Diagnosis of major depressive disorder (MDD), single or recurrent, with a current Major depression episode as diagnosed by the Mini-international Neuropsychiatric Interview (MINI 6.0)
3. Montgomery Asberg Depression Scale score greater than or equal to 15 at baseline.
4. Evidence of decreased executive function as evidenced by either of the following conditions: a) scoring below the mean normative scaled score on the average of the NIH Toolbox executive function measures: Flanker inhibitory control and attention test and the Dimensional sort card test, approximate score 70 - 100 as per PI discretion. b) Discrepancy of at least 10 points between the average of the picture vocabulary score and the reading recognition test score and the average of the Flanker inhibitory control and dimensional card sort test score. c) Frontal Systems Behavior Scale (FRSBE) T scores above 60 (indicative of borderline to clinically significant impairment) and at least 10 points (1 Standard Deviation) above subject's premorbid (pre-depression) scores.

Exclusion Criteria:

1. Inability to complete NIH tool box cognitive testing
2. Inability to provide informed consent
3. <22 score on the Montreal Cognitive Assessment MoCA indicative of moderate to severe cognitive impairment per PI discretion
4. Lifetime diagnosis of bipolar I or II disorder or psychotic disorder as per the MINI interview
5. current psychotic symptoms
6. alcohol or other substance use disorder per DSM V criteria in the past 6 months
7. High risk for suicide (active suicidal ideation/intent or plan and patient is unsafe to be in the outpatient setting), an urgent psychiatric referral will be made in those cases
8. Have a diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), assessed by a study investigator to be primary
9. Previous history of TMS
10. history of failure to an adequate course of electroconvulsive therapy (ECT) such as equal or more than 7-9 electroconvulsive therapy treatments, per PI discretion
11. Major unstable medical illness including advanced/uncontrolled diabetes, hypertension, renal disease or advanced cancer, per PI discretion
12. Psychotropic use other than antidepressants (e.g., Benzodiazepines [more than 2mg of lorazepam equivalent daily], anticonvulsants [except low dose of Neurontin approximately 600mg/day] or cognitive enhancers such as N-Methyl D - Aspartate (NDMA) receptor antagonists [Memantine HCL], psychostimulants [such as methylphenidate or modafinil]) per PI discretion
13. Recent changes or initiation of antidepressant therapy approximately in the last 4 weeks prior to intervention delivery, per PI discretion
14. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
15. contraindications for TMS including the presence of metallic objects within 30 cm of the TMS coil, intracranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed; presence of intracardiac lines, defibrillators or a cardiac pacemaker and unable to assess safety; presence of implanted electronic devices that control physiologic functions and unable to assess safety
16. have a personal history of a primary seizure disorder or a seizure associated with an intracranial lesion
17. History of severe head trauma or neurological disorders that substantially increase seizure risk, per PI discretion
18. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Cristancho, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Washington University in St. Louis School of Medicine - Healthy Mind Lab, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be available upon request to be shared with other researchers interested in geriatric depression and resting state functional connectivity analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication pf study results
Access Criteria: to request information e-mail PI: Pilar Cristancho at cristanchopimiento.l@wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Active iTBS Treatment: Intermittent theta burst stimulation to the dorsolateral prefrontal cortex
  Intermittent Theta Burst Stimulation: Intermittent theta burst stimulation delivered to the dorsolateral prefrontal cortex on the left and right sides of the brain.
- Sham Stimulation: Sham stimulation to the dorsolateral prefrontal cortex.
  Intermittent Theta Burst Stimulation: Intermittent theta burst stimulation delivered to the dorsolateral prefrontal cortex on the left and right sides of the brain.
Period: Overall Study
Arm/Group | Active iTBS Treatment | Sham Stimulation
Started | 10 | 9
Completed | 8 | 9
Not Completed | 2 | 0
Not completed — discontinued study | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active iTBS Treatment | Sham Stimulation | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (5) | 67 (5) | 67 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Montgomery Asberg Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Depression measure
  units on a scale | 23.75 (5.52) | 20.88 (3.88) | 22.23 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Scores From Baseline to the End of the Intervention
Description: We will assess the efficacy of iTBS in improving mood by determining if older adults randomized to iTBS will show significant decreases in the Montgomery-Asberg Depression Rating Scale consistent with improvement of depressive symptoms. The total score for the scale will be reported. The total scores range is 0 - 60 with 0 = minimum score and 60 the maximum score. A low score is better as it denotes less depressive symptoms.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS Treatment | Sham Stimulation
Number analyzed (Participants) | 8 | 9
score on a scale | 10.25 (6.40) | 13.33 (3.70)

2. Primary Outcome: Change in the NIH Toolbox Executive Domain Measure Flanker Inhibitory Control and Attention Test
Description: Improvement in executive function in participants will be assessed by determining if subjects randomized to iTBS show significant increases in their NIH Toolbox Flanker Inhibitory control and attention test from baseline to the end of 6 weeks, compared to those randomized to sham.
  NIH Tool box Flanker inhibitory control and attention test is a validated instrument measuring attention and inhibitory control.
  The age corrected standard score is used, for which the normative mean is 100 and the standard deviation is 15. This score compares the score of the test taker to those in the NIH tool box nationally representative sample at the same age, where a score of 100 indicates performance that was at the national average for the test-taking participant's age. A score of 115 or 85 for example would indicate that the participant's performance is 1SD above or below the national average respectively, when compared with like-aged participants. Higher scores indicate higher performance.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS Treatment | Sham Stimulation
Number analyzed (Participants) | 8 | 9
score on a scale | 1.38 (8.7) | 0.78 (7.42)

3. Primary Outcome: Change in the NIH Tool Box Executive Measure Dimensional Change Card Sort Test
Description: Improvement in executive function in participants will be assessed by determining if subjects randomized to iTBS show significant increases in their NIH Toolbox Dimensional change card sort test from baseline to the end of 6 weeks, compared to those randomized to sham.
  NIH Tool box Dimensional change card sort test is a validated instrument measuring cognitive flexibility.
  The age corrected standard score is used, for which the normative mean is 100 and the standard deviation is 15. This score compares the score of the test taker to those in the NIH tool box nationally representative sample at the same age, where a score of 100 indicates performance that was at the national average for the test-taking participant's age. A score of 115 or 85 for example would indicate that the participant's performance is 1SD above or below the national average respectively, when compared with like-aged participants. Higher scores indicate higher performance.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS Treatment | Sham Stimulation
Number analyzed (Participants) | 8 | 9
score on a scale | 1.00 (10.98) | -1.67 (11.02)

4. Primary Outcome: Change in the NIH Tool Box List Sorting Working Memory Measure
Description: Improvement in executive function in participants will be assessed by determining if subjects randomized to iTBS show significant increases in their NIH Toolbox list sorting working memory test from baseline to the end of 6 weeks, compared to those randomized to sham.
  NIH Tool box list sorting working memory test is a validated instrument measuring working memory.
  The age corrected standard score is used, for which the normative mean is 100 and the standard deviation is 15. This score compares the score of the test taker to those in the NIH tool box nationally representative sample at the same age, where a score of 100 indicates performance that was at the national average for the test-taking participant's age. A score of 115 or 85 for example would indicate that the participant's performance is 1SD above or below the national average respectively, when compared with like-aged participants. Higher scores indicate higher performance.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active iTBS Treatment | Sham Stimulation
Number analyzed (Participants) | 8 | 9
score on a scale | -0.88 (10.77) | -7.00 (14.22)

5. Primary Outcome: Connectivity Change Within the CNN, Fronto-parietal Network
Description: We will test the effects of iTBS on functional connectivity within the CNN ( fronto-parietal network) in depressed older adults obtained using resting state fMRI measuring BOLD signal in the brain.
  Depressed older adults randomized to iTBS versus sham will have a significant increase in functional connectivity within the fronto-parietal network from baseline to week 6.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Active iTBS Treatment | Sham Stimulation
Number analyzed (Participants) | 8 | 9
correlation coefficient | 0.0059 (0.0295) | 0.0153 (0.0347)

6. Primary Outcome: Connectivity Change Within the CNN, Cingulo Opercular Network
Description: We will test the effects of iTBS on functional connectivity within the CNN cingulo opercular network in depressed older adults obtained using resting state fMRI measuring bold signal in the brain.
  Depressed older adults randomized to iTBS versus sham will have a significant increase in functional connectivity within the cingulo-opercular network from baseline to week 6.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Active iTBS Treatment | Sham Stimulation
Number analyzed (Participants) | 8 | 9
correlation coefficient | -0.0070 (0.0329) | 0.0076 (0.0578)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events from baseline (pre-intervention) to the end of of six weeks of the intervention.
Arm/Group | Active iTBS Treatment | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03745768/Prot_SAP_001.pdf